CLINICAL TRIAL: NCT00004644
Title: Phase I/II Study of High-Dose Acyclovir for Central Nervous System or Disseminated Neonatal Herpes Simplex Virus Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/11690; NIAID-17116
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-03

CONDITIONS: Herpes Simplex
Keywords: herpes simplex virus infection; herpesvirus infection; immunologic disorders and infectious disorders; rare disease; viral infection
MeSH Terms: conditions — Herpes Simplex; Herpesviridae Infections; Immune System Diseases; Communicable Diseases; Rare Diseases; Virus Diseases | interventions — Acyclovir

INTERVENTIONS:
Drug: acyclovir

SUMMARY:
OBJECTIVES: I. Evaluate whether high-dose acyclovir decreases acute and long-term morbidity and mortality in neonates with central nervous system or disseminated herpes simplex virus (HSV) infection.

II. Evaluate whether high-dose acyclovir is safe and tolerated in the newborn. III. Assess resistance to antiviral medication. IV. Amplify disease classification for the purpose of predicting prognosis. V. Assess any changes in viral excretion patterns. VI. Evaluate whether antigens and antibodies specific for HSV glycoproteins within the cerebrospinal fluid (CSF) predict long-term neurologic outcome.

VII. Evaluate whether specific antigens and antibodies in the CSF appear late after treatment and are indicative of insidious reactivation of virus in the brain.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Neonates are treated with intravenous acyclovir for 21 days. Patients are followed at day 28, and at 6, 12, 24, 36, and 48 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Herpes simplex virus infection that is disseminated or localized to the central nervous system Virologically confirmed by 1 of the following methods:

* Tissue culture
* Monoclonal antibody staining
* Electron microscopy

--Prior/Concurrent Therapy--

No concurrent antiviral therapy

--Patient Characteristics--

Life expectancy: No imminent demise

Birth weight at least 1200 g Gestational age over 32 weeks

Ages: 0 Years to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25
Dates: Start 1995-02

CONTACTS AND LOCATIONS:
Overall Officials: Richard J. Whitley, Study Chair